CLINICAL TRIAL: NCT01950585
Title: Hydroxyurea in Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130203; 13-H-0203
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-10-23

CONDITIONS: Pulmonary Hypertension
Keywords: Hydroxyurea; Pulmonary Hypertension; Idiopathic Pulmonary Arterial Hypertension; Familial Pulmonary Arterial Hypertension; CD34 + Cells
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension | interventions — Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea

SUMMARY:
Pulmonary arterial hypertension (PAH) is a serious and eventually fatal disease damaging the lungs and the heart. It results from narrowing and eventual blockage of small blood vessels in the lung, due to abnormal proliferation of cells in the blood vessel (arterial). Patients with PAH suffer from fatigue, shortness of breath, low oxygen levels, blood clots and heart failure. No therapies reverse the disease process in the lung arteries, however there are three approved drugs that can temporarily dilate the vessels and improve symptoms. However, all three drugs have significant side effects and toxicities, they do not work effectively in many patients, survival remains on average only 2 to 3 years once symptoms begin, and none of these drugs prevent the underlying disease process in the small arteries of the lung.

PAH is known to develop in patients with a pre-existing class of bone marrow diseases called myeloproliferative disorders (MPDs). We and others have recently shown that patients with PAH have bone marrow changes similar to those seen in patients with MPDs, even without other signs and symptoms of those bone marrow diseases such as anemia or high platelet and white blood cell counts. Compared to healthy volunteers, patients with PAH have a higher frequency of immature stem and progenitor cells able to produce blood cells and vascular wall cells in their bone marrow. They also have higher circulating numbers of these cells in the blood, and increased localization of these cells in the lung blood vessels. When immature bone marrow cells from PAH patients and normal volunteers were infused into mice, the mice receiving PAH marrow cells developed similar lung and heart problems to PAH patients, suggesting that the bone marrow problem is a primary cause of the lung problems, and that the increased numbers of immature bone marrow cells in the bone marrow and blood of PAH patients causes the lung blood vessel disease.

The drug hydroxyurea is used to inhibit the abnormally high level of bone marrow cell proliferation in patients with MPDs. It has been shown to reduce the numbers of circulating immature bone marrow cells in patients with MPDs. Hydroxyurea has been available for almost fifty years, and has been used to treat patients with MPDs, sickle cell anemia, and congenital heart disease for very prolonged periods of time, up to twenty or more years in individual patients. It has an excellent long-term safety profile and few side effects and is generally well tolerated. It does not appear to result in an increased rate of leukemia even with many years of treatment.

In the current protocol, we hypothesize that treating patients with PAH with hydroxyurea will decrease the level of circulating immature bone marrow cells and interrupt the abnormal narrowing and occlusion of lung arteries. We will treat patients with moderately severe primary (no known underlying cause) PAH with 6 months of hydroxyurea, carefully monitoring side effects and adjusting dosage as necessary, and measure the effect on circulating immature cells, lung blood vessel pressures, other blood markers of active PAH, and exercise tolerance.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a serious and eventually fatal disease damaging the lungs and the heart. It results from narrowing and eventual blockage of small blood vessels in the lung, due to abnormal proliferation of cells in the blood vessel (arterial). Patients with PAH suffer from fatigue, shortness of breath, low oxygen levels, blood clots and heart failure. No therapies reverse the disease process in the lung arteries, however there are three approved drugs that can temporarily dilate the vessels and improve symptoms. However, all three drugs have significant side effects and toxicities, they do not work effectively in many patients, survival remains on average only 2 to 3 years once symptoms begin, and none of these drugs prevent the underlying disease process in the small arteries of the lung.

PAH is known to develop in patients with a pre-existing class of bone marrow diseases called myeloproliferative disorders (MPDs). We and others have recently shown that patients with PAH have bone marrow changes similar to those seen in patients with MPDs, even without other signs and symptoms of those bone marrow diseases such as anemia or high platelet and white blood cell counts. Compared to healthy volunteers, patients with PAH have a higher frequency of immature stem and progenitor cells able to produce blood cells and vascular wall cells in their bone marrow. They also have higher circulating numbers of these cells in the blood, and increased localization of these cells in the lung blood vessels. When immature bone marrow cells from PAH patients and normal volunteers were infused into mice, the mice receiving PAH marrow cells developed similar lung and heart problems to PAH patients, suggesting that the bone marrow problem is a primary cause of the lung problems, and that the increased numbers of immature bone marrow cells in the bone marrow and blood of PAH patients causes the lung blood vessel disease.

The drug hydroxyurea is used to inhibit the abnormally high level of bone marrow cell proliferation in patients with MPDs. It has been shown to reduce the numbers of circulating immature bone marrow cells in patients with MPDs. Hydroxyurea has been available for almost fifty years, and has been used to treat patients with MPDs, sickle cell anemia, and congenital heart disease for very prolonged periods of time, up to twenty or more years in individual patients. It has an excellent long-term safety profile and few side effects and is generally well tolerated. It does not appear to result in an increased rate of leukemia even with many years of treatment.

In the current protocol, we hypothesize that treating patients with PAH with hydroxyurea will decrease the level of circulating immature bone marrow cells and interrupt the abnormal narrowing and occlusion of lung arteries. We will treat patients with moderately severe primary (no known underlying cause) PAH with 6 months of hydroxyurea, carefully monitoring side effects and adjusting dosage as necessary, and measure the effect on circulating immature cells, lung blood vessel pressures, other blood markers of active PAH, and exercise tolerance.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old
* Patients with idiopathic or familial PAH with WHO II-III performance status
* On PAH medications that have not changed and are stable for the past two months
* Seronegative for HIV antibody, hepatitis B antigen, and hepatitis C antibody.

EXCLUSION CRITERIA:

* Thrombocytopenia with platelets less than 100,000/mm3, anemia with hemoglobin less than 10.5g/dL or neutropenia with ANC less than 1500/mm3
* Creatinine > 2.0mg/dL
* Hepatic insufficiency (transaminase levels >4 fold the upper limit of normal or bilirubin >2 fold the upper limit of normal)
* Severe arterial hypertension (systolic blood pressure >200mmHg or diastolic >120mmHg)
* Female subjects who are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
* Participation in any other investigative treatment studies at the time of enrollment
* Unable to understand the investigational nature of the study or give informed consent (i.e. decisionally impaired)<TAB>
* Evidence of major bleeding or active infection
* Known allergy to the study drug or drugs similar to the study drug
* Subjects with known liver cirrhosis or chronic active hepatitis.
* HIV positivity
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 30 days is likely
* Presence of 9;22 BCR/ABL translocation as detected by conventional bone marrow cytogenetics or PCR for BCR/ABL transcript, or presence of JAK2 V617F mutation in bone marrow or peripheral blood cells.
* On beta-blocker therapy requiring dose adjustment.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09-06; Primary Completion 2014-10-23 (Actual); Study Completion 2014-10-23 (Actual)

PRIMARY OUTCOMES:
The change in concentration of CD34+ circulating progenitors from baseline to 6 months (24 weeks (+/- 7 days)) on hydroxyurea. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Moonjung Jung, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)

REFERENCES:
- [Background] Masri FA, Xu W, Comhair SA, Asosingh K, Koo M, Vasanji A, Drazba J, Anand-Apte B, Erzurum SC. Hyperproliferative apoptosis-resistant endothelial cells in idiopathic pulmonary arterial hypertension. Am J Physiol Lung Cell Mol Physiol. 2007 Sep;293(3):L548-54. doi: 10.1152/ajplung.00428.2006. Epub 2007 May 25. PMID 17526595
- [Background] Farha S, Asosingh K, Xu W, Sharp J, George D, Comhair S, Park M, Tang WH, Loyd JE, Theil K, Tubbs R, Hsi E, Lichtin A, Erzurum SC. Hypoxia-inducible factors in human pulmonary arterial hypertension: a link to the intrinsic myeloid abnormalities. Blood. 2011 Mar 31;117(13):3485-93. doi: 10.1182/blood-2010-09-306357. Epub 2011 Jan 21. PMID 21258008
- [Background] Asosingh K, Farha S, Lichtin A, Graham B, George D, Aldred M, Hazen SL, Loyd J, Tuder R, Erzurum SC. Pulmonary vascular disease in mice xenografted with human BM progenitors from patients with pulmonary arterial hypertension. Blood. 2012 Aug 9;120(6):1218-27. doi: 10.1182/blood-2012-03-419275. Epub 2012 Jun 28. PMID 22745307